CLINICAL TRIAL: NCT05594550
Title: Evaluation of the Prognostic Value of T7 and T12 Slices on Mortality in Resuscitation Patients With ARDS Caused by SARS-COV2 Infection
Acronym: MUSCOV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: NGUYEN 2022
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Acute Respiratory Distress Syndrom (SARS-Cov 2)
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 28-day survival: Alive 28 days after intensive care admission
  Interventions: Other: Data collection; Other: analysis of thoracic scans
- 28-day death: Deceased 28 days after intensive care admission
  Interventions: Other: Data collection; Other: analysis of thoracic scans

INTERVENTIONS:
Other: Data collection — Demographic data:
  Age, Sex, weight, height, main history and treatments.
  - Biological data: CRP, PCT, albumin, pre-albumin
Other: analysis of thoracic scans — muscle area calculated on the T7 and T12 thoracic slices

SUMMARY:
Sarcopenia is a risk factor for adverse outcome in critically ill patients. Sarcopenia might be estimated from muscle surface measure on tomodensitometry.

The purpose of the study is to identify if muscle surfaces measured on thoracic tomodensitometry are associated with mortality in patients with acute respiratory distress syndrome due to SARS-Cov-2.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in intensive care for SARS-Cov-2 infection since january 2020
* Thoracic TDM within the 30 day preceding ICU admission and up to 24 hours after ICU admission

Exclusion Criteria:

* Pregnancy
* Neuromuscular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with acute respiratory syndrome due to SARS-Cov-2
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
measurement of muscle area at T7 level indexed in cm²/m². | At hospital admission
  use of CT measurements to discriminate between the 2 groups (deceased versus alive)

SECONDARY OUTCOMES:
Duration of mechanical ventilation | within the 28 days
Ventilator free days | within the 28 days
number of days in Intensive care unit | within the 28 days
number of days in hospital | within the 28 days